CLINICAL TRIAL: NCT04156594
Title: Preoperative Self-assessment for Cardio-pulmonary Risk Stratification
Acronym: PRESELECT
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, André Dankert, MD, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: PV7061
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Lung Diseases, Obstructive; Postoperative Complications; Cardiac Event
Keywords: self-assessment; post operative pulmonary complication; ExerciseTest
MeSH Terms: conditions — Lung Diseases, Obstructive; Postoperative Complications; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective study intends to development and validation a patient self-assessment questionnaire. The aim of the self-assessment, by questionnaire, is to estimate the risk of postoperative pulmonary complications (PPC).

DETAILED DESCRIPTION:
PPC are common adverse events operative patients. Existing concepts of pulmonary risk evaluation are based on complex risk scores, preoperative apparatus examinations, laboratory parameters and medical findings. The significance of apparatus diagnostics for the preoperative Pulmonary risk evaluation is highly controversial and guidelines recommend a reluctant use. A large prospective study (PREDICT, unpublished to date, NCT02566343) showed that lung function assessment in patients with COPD symptoms undergoing major non-cardiac surgery did not improve the anamnestic risk assessment. In a large study it could be shown that a subjective self-assessment of physical performance by means of a structured questionnaire (DASI), in contrast to a subjective medical assessment, suitable for predicting perioperative cardiac events. Our unpublished data show that a subjective self-assessment of "limited exercise capacity" in patients with COPD is predictive of PPC is suitable.

Objectives:

* Development of a self-assessment questionnaire as part of a Delphi trial
* Validation of the self-assessment questionnaire

Methodology:

Prospective observational, case control study of 5000 patients undergoing surgery in general anesthesia (estimated enrollment of 5500 patients with a dropout rate of approximately 10%).

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Operations in general anesthesia

Exclusion Criteria:

* < 18 Years
* Pregnancy
* Lack of cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for operations in general anesthesia, who present in the pre-assessment clinic of the University Medical Center Hamburg-Eppendorf during the study recruitment period, will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 5500 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Postoperative pulmonary complications (PPC) | until hospital discharge up to 6 months after surgery
  European Perioperative Clinical Outcome (EPCO) definitions

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | until hospital discharge up to 6 months after surgery
  European Perioperative Clinical Outcome (EPCO) definitions
New diagnoses in the context of the current hospital stay New pulmonary or cardiac diagnoses | until hospital discharge up to 6 months after surgery
  New diagnoses in the context of the current hospital stay New pulmonary or cardiac diagnoses
Duration of hospitalization (days) | until hospital discharge up to 6 months after surgery
  Duration of hospitalization (days)
in-hospital mortality | until hospital discharge up to 6 months after surgery
  in-hospital mortality
Length of stay in the intensive care unit (days) | until hospital discharge up to 6 months after surgery
  Length of stay in the intensive care unit (days)

CONTACTS AND LOCATIONS:
Overall Officials: André Dankert, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Background] Gupta H, Ramanan B, Gupta PK, Fang X, Polich A, Modrykamien A, Schuller D, Morrow LE. Impact of COPD on postoperative outcomes: results from a national database. Chest. 2013 Jun;143(6):1599-1606. doi: 10.1378/chest.12-1499. PMID 23287892
- [Background] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504
- [Background] Vogelmeier CF, Criner GJ, Martinez FJ, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Chen R, Decramer M, Fabbri LM, Frith P, Halpin DM, Lopez Varela MV, Nishimura M, Roche N, Rodriguez-Roisin R, Sin DD, Singh D, Stockley R, Vestbo J, Wedzicha JA, Agusti A. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report: GOLD Executive Summary. Eur Respir J. 2017 Mar 6;49(3):1700214. doi: 10.1183/13993003.00214-2017. Print 2017 Mar. PMID 28182564
- [Background] Wijeysundera DN, Pearse RM, Shulman MA, Abbott TEF, Torres E, Ambosta A, Croal BL, Granton JT, Thorpe KE, Grocott MPW, Farrington C, Myles PS, Cuthbertson BH; METS study investigators. Assessment of functional capacity before major non-cardiac surgery: an international, prospective cohort study. Lancet. 2018 Jun 30;391(10140):2631-2640. doi: 10.1016/S0140-6736(18)31131-0. PMID 30070222